CLINICAL TRIAL: NCT00731809
Title: Evaluation of PET CT in the Management of Patients With Crohn's Disease.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Hanna Brrnstine MD, Beilinson Hospital Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 004945
Record Dates: First submitted 2008-08-03; First posted 2008-08-11 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): PET CT
  Interventions: Radiation: FDG PET CT

INTERVENTIONS:
Radiation: FDG PET CT — FDG PET CT

SUMMARY:
18F-FDG PET/CT (2-[fluorine-18] fluoro-2-deoxy-D-glucose, Positron emission tomography- CT) is a noninvasive technique that allows quantifying and precisely localizing 18F-FDG uptake in the entire body. 18F-FDG uptake is caused by increased local metabolic activity. Such increased uptake has been described not only in neoplastic lesions but also in inflammatory lesions. In this condition, uptake has been correlated with local stimulation of tumor necrosis factor, and with monocyte priming and activation. A physiologic variable uptake may be observed in the bowel, especially the cecum, and has limited the use of PET in inflammatory bowel diseases. The advantage of combined PET and CT devices lead to significant improvements in the interpretation of the bowel areas, and greatly reduces the number of false-positive findings in the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspicious for active disease:

  * Patients with suspected but undiagnosed Crohn's disease
  * Patients with serological markers of inflammation (elevated ESR, CRP or thrombocytosis) but clinically in remission
  * Patients with a stricture which might be fibrous in which case surgery is indicated or inflammatory for which medical management is indicated
  * Able to sign a consent form

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Infectious colitis determined at the initial checkup
* Allergy to iodine contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel